CLINICAL TRIAL: NCT00001724
Title: Evaluation of the Analgesic Effects of Locally Applied Flurbiprofen and Bupivacaine in the Oral Surgery Model
Brief Title: Local Flurbiprofen to Treat Pain Following Wisdom Tooth Extraction
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 980035; 98-D-0035
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2008-03-04 (Estimated); Status verified 2001-11

CONDITIONS: Pain
Keywords: Pain; Microencapsulated Drug; NSAID; Acute Inflammation; Peripheral Administration; Dose-Response; Relative Potency Assay; Pharmacokinetics
MeSH Terms: conditions — Pain | interventions — Flurbiprofen

INTERVENTIONS:
Drug: Flurbiprofen

SUMMARY:
This study will evaluate the effectiveness of the non-steroidal anti-inflammatory drug flurbiprofen (Ansaid® (Registered Trademark)) in relieving pain following oral surgery. Flurbiprofen is approved by the Food and Drug Administration for treatment of arthritis pain.

Patients 16 years of age and older requiring third molar (wisdom tooth) extraction may be eligible for this study.

Patients will undergo oral surgery to remove two lower third molar teeth. Before surgery, they will be given a local anesthetic (lidocaine with epinephrine) injected in the mouth and a sedative (Versed) infused through a catheter (thin plastic tube) placed in an arm vein. At the time of surgery, patients will also be given flurbiprofen or a placebo formulation (look-alike substance with no active ingredient) directly into the extraction site and a capsule that also may contain flurbiprofen or placebo. One in seven patients will receive only placebo.

All patients will fill out pain questionnaires and stay in the clinic for up to 6 hours for observation of bleeding and medication side effects. Patients who do not have satisfactory pain relief from the test medicine after surgery may request a standard pain reliever. A small blood sample will be collected during surgery and at 15 minutes, one-half hour and 1, 2, 3, 4, 5, 6, 24 and 48 hours after surgery to measure flurbiprofen blood levels. A total of 33 ml (about 2 tablespoons) of blood will be drawn for these tests. Samples collected on the day of surgery will be drawn from the catheter used to administer the sedative; the 24- and 48-hour samples will be taken by needle from an arm or hand vein. Urine samples will also be collected between 4 and 6 hours after surgery and again at 24 and 48 hours after surgery.

DETAILED DESCRIPTION:
This study proposes to evaluate the analgesic efficacy, tissue response, and adverse effects of microencapsulated preparations of a nonsteroidal anti-inflammatory drug (NSAID) and a long-acting local anesthetic administered into post-extraction sites prior to pain onset. Subjects (N=84) will have two mandibular impacted third molars removed and be randomly allocated to receive one of six possible treatments placed into the sockets: 0 mg (placebo formulation), 3.125 mg, 6.25 mg, 12.5 mg, or 25 mg flurbiprofen, or 50 mg bupivacaine. Each patient in these six groups (N=12/group) will also receive an oral placebo capsule. The seventh group of subjects will receive a placebo at the extraction sites and 25 mg of flurbiprofen orally. Subjects will remain at the clinic for six hours following drug administration to record every 30 minutes the offset of mandibular anesthesia, postoperative pain intensity, side effects, and for observation of recurrent bleeding. Demonstration of a dose-responsive relationship for flurbiprofen at doses lower than needed for analgesia following oral administration will provide the basis for a second study in which an optimal dose of flurbiprofen will be combined with bupivacaine.

ELIGIBILITY:
Patients of either sex requiring removal of two impacted mandibular third molars (partial bony or soft tissue impaction).

16 years of age of older.

Indicates willingness to undergo oral surgery with local anesthesia and intravenous midazolam only.

Willing to return for the removal of the remaining maxillary third molars at a second appointment.

Patients with a history of allergy to flurbiprofen, aspirin, or any NSAID will be excluded.

Those with a history of aspirin or NSAID-induced asthma will be excluded.

Females of childbearing potential who are not practicing adequate contraception will be excluded.

Pregnant or nursing females will be excluded.

Patients with recent history or present signs of renal, hepatic, endocrine, pulmonary, cardiac, gastrointestinal, neurologic, or cerebral function impairment will be excluded.

Those with psychiatric disorders will be excluded.

Patients who have taken an investigational drug within 30 days of this study will be excluded.

Those who have taken another analgesic, steroid, opioid, or NSAID within 24 hours prior to the study will be excluded.

Those with an absence of bilateral local anesthesia during surgery as evidenced by anesthesia or paresthesia of the lower lip postoperatively will be excluded.

Patients who use drugs which will interact with NSAID such as aspirin, warfarin, probenecid, methotrexate, lithium and diuretics will be excluded.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100
Dates: Start 1997-11; Study Completion 2001-11

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Dental And Craniofacial Research (NIDCR), Bethesda, Maryland, United States

REFERENCES:
- [Background] Dionne RA. Suppression of dental pain by the preoperative administration of flurbiprofen. Am J Med. 1986 Mar 24;80(3A):41-9. doi: 10.1016/0002-9343(86)90110-5. PMID 3515923
- [Background] Moore UJ, Seymour RA, Rawlins MD. The efficacy of locally applied aspirin and acetaminophen in postoperative pain after third molar surgery. Clin Pharmacol Ther. 1992 Sep;52(3):292-6. doi: 10.1038/clpt.1992.144. PMID 1526087
- [Background] Allison MC, Howatson AG, Torrance CJ, Lee FD, Russell RI. Gastrointestinal damage associated with the use of nonsteroidal antiinflammatory drugs. N Engl J Med. 1992 Sep 10;327(11):749-54. doi: 10.1056/NEJM199209103271101. PMID 1501650